CLINICAL TRIAL: NCT02449473
Title: A Multicentre, Randomized, Double-blind, Parallel Group, Placebo Controlled, 12-Week, Ph 2 Study to Evaluate the Effect of Tralokinumab on Airway Inflammation in Adults With Asthma Inadequately Controlled on Inhaled Corticosteroid (MESOS)
Brief Title: Study to Evaluate Efficacy & Safety of Tralokinumab in Subjects With Asthma Inadequately Controlled on Corticosteroids
Acronym: MESOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D2210C00014
Record Dates: First submitted 2015-05-18; First posted 2015-05-20 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Asthma
Keywords: Asthma; Reactive Airways; Respiratory Tract Disease; Obstructive Tract Disease; Lung Diseases
MeSH Terms: conditions — Asthma; Respiratory Tract Diseases; Lung Diseases | interventions — tralokinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tralokinumab Dose Regimen (Experimental): Tralokinumab Subcutaneous Injection
  Interventions: Biological: Tralokinumab
- Placebo Dose Regimen (Placebo Comparator): Placebo Subcutaneous Injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Tralokinumab — Subcutaneous Injection
  Arms: Tralokinumab Dose Regimen
Other: Placebo — Subcutaneous Injection
  Arms: Placebo Dose Regimen

SUMMARY:
A Multicentre, Randomized, Double-blind, Parallel Group, Placebo Controlled, 12-Week, Phase 2 Study to Evaluate the Effect of Tralokinumab on Airway Inflammation in Adults with Asthma Inadequately Controlled on Inhaled Corticosteroid.

DETAILED DESCRIPTION:
This is a multicentre, randomized, double-blind, parallel group, placebo-controlled, phase 2 study to designed evaluate the effect of a 300 mg dose of tralokinumab administered subcutaneously every 2 weeks on airway inflammation in adults with asthma inadequately controlled on inhaled corticosteroids (ICS) with or without other controllers. Approximately 80 subjects will be randomized. Subjects will receive tralokinumab, or placebo, administered via subcutaneous injection at the study site, over a 12 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years
2. Documented physician-diagnosed asthma for at least 12 months prior to enrolment (v1)
3. Documented treatment with an asthma controller regimen requiring treatment with ICS (minimum dose of ≥ 250 ug fluticasone propionate via dry powder inhaler equivalents total daily dose) alone or in combination ≥ 6 months and that has been taken at a stable dose for at least 1 month prior to enrolment (v1)
4. Additional maintenance asthma controller medications must be given at a stable dose for at least 1 month prior to v1.
5. At enrolment (v1) the subject must have a predicted normal value (PNV) for the pre-bronchodilator (BD) FEV1>50% and more than 1L.
6. Post-BD reversibility in FEV1 of ≥12% and ≥200 mL at enrolment (v1).

Exclusion Criteria:

1. History of interstitial lung disease, chronic obstructive pulmonary disease (COPD), or other clinically significant lung disease other than asthma.
2. History of anaphylaxis following any biologic therapy.
3. Hepatitis B, C or HIV
4. Pregnant or breastfeeding
5. History of cancer
6. Current tobacco smoking or a history of tobacco smoking for >10 pack-years.
7. Previous receipt of tralokinumab

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Brightling, MD, Principal Investigator — Institute for Lung Health, United Kingdom
Locations (15):
- Canada (3):
  - Research Site, Vancouver, British Columbia
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Denmark (5):
  - Research Site, Aalborg
  - Research Site, Århus C
  - Research Site, Hvidovre
  - Research Site, København NV
  - Research Site, Odense C
- United Kingdom (7):
  - Research Site, Belfast
  - Research Site, Glasgow
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Nottingham
  - Research Site, Southampton

REFERENCES:
- [Derived] Diver S, Sridhar S, Khalfaoui LC, Russell RJ, Emson C, Griffiths JM, de Los Reyes M, Yin D, Colice G, Brightling CE. Feno differentiates epithelial gene expression clusters: Exploratory analysis from the MESOS randomized controlled trial. J Allergy Clin Immunol. 2022 Oct;150(4):830-840. doi: 10.1016/j.jaci.2022.04.024. Epub 2022 May 7. PMID 35537502
- [Derived] Russell RJ, Chachi L, FitzGerald JM, Backer V, Olivenstein R, Titlestad IL, Ulrik CS, Harrison T, Singh D, Chaudhuri R, Leaker B, McGarvey L, Siddiqui S, Wang M, Braddock M, Nordenmark LH, Cohen D, Parikh H, Colice G, Brightling CE; MESOS study investigators. Effect of tralokinumab, an interleukin-13 neutralising monoclonal antibody, on eosinophilic airway inflammation in uncontrolled moderate-to-severe asthma (MESOS): a multicentre, double-blind, randomised, placebo-controlled phase 2 trial. Lancet Respir Med. 2018 Jul;6(7):499-510. doi: 10.1016/S2213-2600(18)30201-7. Epub 2018 May 21. PMID 29793857
- [Derived] Panettieri RA Jr, Wang M, Braddock M, Bowen K, Colice G. Tralokinumab for the treatment of severe, uncontrolled asthma: the ATMOSPHERE clinical development program. Immunotherapy. 2018 Mar 1;10(6):473-490. doi: 10.2217/imt-2017-0191. Epub 2018 Mar 14. PMID 29536781
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3064&filename=d2210c00014-sap-redacted2019.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3064&filename=d2210c00014-csp-Redacted2019.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 29 Sep 2015; Last patient last visit: 21 Jun 2017. Study performed at 14 sites in 3 countries. Patients maintained on currently prescribed inhaled corticosteroid (≥250 micrograms fluticasone dry powder formulation equivalents total daily dose) + any additional maintenance asthma controller medication throughout the study.
Pre-assignment Details: 79 patients were randomised to receive investigational product (IP) and all those randomised received treatment.
Groups:
- Tralo 300 mg Q2W: Tralokinumab 300 milligrams (mg) administered subcutaneously every 2 weeks (Q2W) over a 12-week treatment period (up to 6 doses).
- Placebo: Placebo administered subcutaneously Q2W over a 12-week treatment period (up to 6 doses).
Period: Overall Study
Arm/Group | Tralo 300 mg Q2W | Placebo
Started | 39 | 40
Completed | 39 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients in the full analysis set (FAS) and who received any IP (tralokinumab or placebo) were included in the baseline analysis.
Groups:
- Tralo 300 mg Q2W: Tralokinumab 300 mg administered subcutaneously Q2W over a 12-week treatment period (up to 6 doses).
- Total: Total of all reporting groups
Arm/Group | Tralo 300 mg Q2W | Placebo | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.1 (14.2) | 50.1 (14.2) | 48.6 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 16 | 20 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 34 | 39 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12, Expressed as a Ratio, in Number of Airway Submucosal Eosinophils
Description: The number of airway submucosal eosinophils per millimetre squared (mm^2) was determined by microscopic evaluation of bronchoscopic biopsies. The ratio of post-randomisation value at Week 12 to baseline value was computed as (Week 12 value / baseline value). The change from baseline to Week 12 (ratio) in the number of airway submucosal eosinophils is presented as geometric mean ± standard deviation (SD) of log values.
Time Frame: Baseline (Week 0) and Week 12
Population: The FAS included all randomised patients who received any IP, irrespective of their protocol adherence and continued participation in the study. Only patients with data available at the timepoints of testing were included in the analyses.
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 35 | 39
Ratio | 1.29 (2.06) | 1.07 (1.87)
Statistical Analysis 1: Comparison: Tralo 300 mg Q2W vs Placebo; Comparison of change from baseline, expressed as a ratio, in airway submucosal eosinophils; Tralo 300 mg Q2W vs placebo. The null hypothesis was that the change in airway submucosal eosinophils at Week 12 on tralokinumab was equal to the corresponding change on placebo; Test type: Superiority — The model included treatment group as fixed effect and baseline log-transformed airway submucosal eosinophils as a continuous covariate. No interaction terms were included in the model. The analysis was performed using log-transformed data. All group comparisons from analysis of covariance (ANCOVA) model were based on Type III sums of squares; p = 0.3862, ANCOVA; Least square (LS) geometric mean ratio = 1.43, 95% CI 2-sided [0.63 to 3.27]

2. Secondary Outcome: Change From Baseline to Week 12, Expressed as a Ratio, in Number of Blood Eosinophils
Description: The blood eosinophil count was obtained from the total and differential white blood cell counts. The ratio of post-randomisation value at Week 12 to baseline value was computed as (Week 12 value / baseline value). The change from baseline to Week 12 (ratio) in the number of blood eosinophils is presented as geometric mean ± SD of log values.
Time Frame: Baseline (Week 0) and Week 12
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 33 | 37
Ratio | 1.10 (0.38) | 0.91 (0.46)
Statistical Analysis 1: Comparison: Tralo 300 mg Q2W vs Placebo; Comparison of change from baseline, expressed as a ratio, in blood eosinophil count; Tralo 300 mg Q2W vs placebo; Test type: Superiority — The repeated measures analysis included treatment group, baseline log-transformed eosinophils and visit as fixed effects. Treatment-by-visit interaction was also included. The analysis was performed using log-transformed data. A restricted maximum likelihood (REML) approach was used. An unstructured variance-covariance matrix was used to model the within-subject errors; p = 0.0546, Repeated measures analysis; LS geometric mean ratio = 1.21, 95% CI 2-sided [1.00 to 1.48]

3. Secondary Outcome: Change From Baseline to Week 12, Expressed as a Ratio, in Number of Differential Sputum Eosinophils
Description: Sputum induction was performed to obtain satisfactory samples of sputum originating from the airways. The ratio of post-randomisation value at Week 12 to baseline value was computed as (Week 12 value / baseline value). The change from baseline to Week 12 (ratio) in the number of eosinophils in induced sputum is presented as geometric mean ± SD of log values.
Time Frame: Baseline (Week 0) and Week 12
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 16 | 17
Ratio | 0.20 (3.16) | 0.47 (3.63)
Statistical Analysis 1: Comparison: Tralo 300 mg Q2W vs Placebo; Comparison of change from baseline, expressed as a ratio, in differential sputum eosinophils; Tralo 300 mg Q2W vs placebo; Test type: Superiority — The repeated measures analysis included treatment group, baseline log-transformed differential sputum eosinophils and visit as fixed effects. Treatment-by-visit interaction was also included. The analysis was performed using log-transformed data. A REML approach was used. An unstructured variance-covariance matrix was used to model the within-subject errors; p = 0.6334, Repeated measures analysis; LS geometric mean ratio = 0.57, 95% CI 2-sided [0.06 to 6.00]

4. Secondary Outcome: Change From Baseline to Week 12, Expressed as a Ratio, in Blood Free Eosinophil Cationic Protein (ECP) Concentrations
Description: ECP concentrations were determined to assess evidence of activation of eosinophils in blood. The ratio of post-randomisation value at Week 12 to baseline value was computed as (Week 12 value / baseline value). The change from baseline to Week 12 (ratio) in blood free ECP concentrations is presented as geometric mean ± SD of log values.
Time Frame: Baseline (Week 0) and Week 12
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 24 | 28
Ratio | 1.07 (0.40) | 0.92 (0.47)
Statistical Analysis 1: Comparison: Tralo 300 mg Q2W vs Placebo; Comparison of change from baseline, expressed as a ratio, in blood free ECP concentration; Tralo 300 mg Q2W vs placebo; Test type: Superiority — The repeated measures analysis included treatment group, baseline log-transformed blood free ECP and visit as fixed effects. Treatment-by-visit interaction was also included. The analysis was performed using log-transformed data. A REML approach was used. An unstructured variance-covariance matrix was used to model the within-subject errors; p = 0.3769, Repeated measures analysis; LS geometric mean ratio = 1.11, 95% CI 2-sided [0.88 to 1.40]

5. Secondary Outcome: Change From Baseline to Week 12, Expressed as a Ratio, in Sputum Free ECP Concentrations
Description: ECP concentrations were determined to assess evidence of activation of eosinophils in sputum. The ratio of post-randomisation value at Week 12 to baseline value was computed as (Week 12 value / baseline value). The change from baseline to Week 12 (ratio) in sputum free ECP concentrations is presented as geometric mean ± SD of log values.
Time Frame: Baseline (Week 0) and Week 12
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Tralo 300 mg Q2W | Placebo
Number analyzed (Participants) | 16 | 17
Ratio | 0.66 (1.21) | 1.83 (1.41)
Statistical Analysis 1: Comparison: Tralo 300 mg Q2W vs Placebo; Comparison of change from baseline, expressed as a ratio, in sputum free ECP concentration; Tralo 300 mg Q2W vs placebo; Test type: Superiority — The repeated measures analysis included treatment group, baseline log-transformed sputum free ECP and visit as fixed effects. Treatment-by-visit interaction was also included. The analysis was performed using log-transformed data. A REML approach was used. An unstructured variance-covariance matrix was used to model the within-subject errors; p = 0.1126, Repeated measures analysis; LS geometric mean ratio = 0.49, 95% CI 2-sided [0.20 to 1.20]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Data is reported for adverse events during the treatment period (onset date ≥ the first day of IP and ≤ the last day of IP + 2 weeks). Patient population was the safety analysis set which included all patients who received any IP, classified according to the treatment they actually received.
Arm/Group | Tralo 300 mg Q2W | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/39 | 1/40
Other Adverse Events (participants affected / at risk) | 30/39 | 27/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tralo 300 mg Q2W (N=39) | Placebo (N=40)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tralo 300 mg Q2W (N=39) | Placebo (N=40)
Viral upper respiratory tract infection (Infections and infestations) | 8 (10) | 17 (20)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 9 (18)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Injection site erythema (General disorders) | 3 (3) | 0 (0)
Injection site pain (General disorders) | 2 (3) | 0 (0)
Injection site pruritus (General disorders) | 2 (3) | 0 (0)
Injection site swelling (General disorders) | 2 (3) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (3)
Weight increased (Investigations) | 2 (2) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The results for differential sputum eosinophils and sputum free ECP levels should be viewed cautiously due to the small sample size and wide variability in results for sputum analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-01-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT02449473/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT02449473/SAP_001.pdf